CLINICAL TRIAL: NCT02901509
Title: Epidémie de Chikungunya à l'île de La Réunion : Effet à Dix Ans de l'Infection Sur la qualité de Vie Dans la Cohorte TELECHIK
Brief Title: Impact of the Chikungunya Outbreak in Reunion Island on the Quality of Life After 10 Years
Acronym: QoLCHIK
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/CHU/QoLCHIK
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Chikungunya Fever; Quality of Life
Keywords: Chikungunya; Quality of Life
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CHIK +: People with chikungunya diagnosis (serodiagnosis)
- CHIK -: People without chikungunya diagnosis (negative serology)

SUMMARY:
QoLCHIK study aims at evaluating impact of chikungunya infection on the quality of life of infected people during the 2005-2006 outbreak in Reunion Island and followed in the TELECHIK cohort by comparing scores of SF-36 health survey.

DETAILED DESCRIPTION:
QoLCHIK is a prospective cohort telephone study on the quality of life of people from the TELECHIK cohort, measured by the SF-36 health survey. TELECHIK was a telephone survey conducted 2 years after the 2005-2006 outbreak in Reunion Island and drawn from the SEROCHIK study which aimed at assessing the seroprevalence of chinkungunya over the island between august and october 2006.

A sample of 440 people (220 per group) was calculated and to be drawn from TELECHIK cohort, 220 with a serodiagnosis of chikungunya and 220 with negative serology.

ELIGIBILITY:
Inclusion Criteria:

* People from the TELECHIK cohort

Exclusion Criteria:

* People with other diseases or disorders which could impact quality of life (predefined list)
* Minor
* Elderly over 85 yo
* People with a risk of exposure (in an endemic/epidemic area) after 2005-2006 Reunion Island outbreak

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: TELECHIK cohort population drawn for telephone survey
Sampling Method: Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2016-06; Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Mean score SF-36 health survey | 1 year

SECONDARY OUTCOMES:
Mean score AQ-5D health survey | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Universitaire de La Réunion, Saint-Pierre, France

IPD SHARING:
Plan to Share IPD: No